CLINICAL TRIAL: NCT00670670
Title: A Prospective, Randomized Clinical Study on the Effects of CPP-ACP Paste on Plaque, Gingivitis and White Spot Lesions in Orthodontic Patients - Part 1
Brief Title: A Prospective, Randomized Clinical Study on the Effects of Casein Phosphopeptide-amorphous Calcium Phosphate (CPP-ACP) Paste on Plaque, Gingivitis and White Spot Lesions in Orthodontic Patients - Part 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: GC Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/187 - Part 1
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Early Caries Lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CPP-ACP (GC Tooth Mousse)
  Interventions: Device: CPP-ACP (GC Tooth Mousse)
- 2 (Experimental): CPP-ACP (GC MI Paste Plus)
  Interventions: Device: CPP-ACP (GC MI Paste Plus)
- 3 (No Intervention): Control group

INTERVENTIONS:
Device: CPP-ACP (GC Tooth Mousse) — Calcium and phosphate
  Arms: 1
Device: CPP-ACP (GC MI Paste Plus) — Calcium, phosphate and fluoride
  Arms: 2

SUMMARY:
Influence of CPP-ACP paste on the evolution and appearance of white spot lesions in orthodontic patients after removal of the fixed appliances.

ELIGIBILITY:
Inclusion Criteria:

* one or more white spot lesion at the time of removal of fixed appliances

Exclusion Criteria:

* white spots already present before start orthodontic treatment

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 325 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2011-01-21 (Actual); Study Completion 2011-04-26 (Actual)

PRIMARY OUTCOMES:
Amelioration of the opacity of white spots into a more natural tooth-like translucency | After 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guy De Pauw, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be